CLINICAL TRIAL: NCT01528761
Title: Prosocial Behavior and Volunteerism to Promote Physical Activity in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00017741; 1R01HL109429-04 (NIH)
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Physical Activity
Keywords: physical activity; older adults; physical function; health-related quality of life; prosocial behavior; social cognitive theory
MeSH Terms: conditions — Motor Activity; Altruism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prosocial Behavior Physical Activity (Experimental): The PBPA condition involves a cognitive-behavioral intervention to teach participants the behavioral skills to engage in independent physical activity. Participants will engage in supervised physical activity delivered two times a week during months 1 to 3 at the William G. White, Jr. Family YMCA in Winston-Salem, NC. During months 4 to 6, supervised sessions will be held once per week, and sessions will be held once per month in months 7 to 9. Participants will engage in completely independent physical activity in months 10 to 12. PBPA participants will also be able to earn boxes of food for donation to the Second Harvest Food Bank (SHFB) of Northwest North Carolina based upon their weekly physical activity. Lowe's Foods, a regional grocery chain, will donate the food. Participants in the PBPA intervention also will receive a 12-month membership to the William G. White, Jr. Family YMCA at no cost.
  Interventions: Behavioral: Prosocial Behavior Physical Activity (PBPA)
- Healthy Aging (HA) (Active Comparator): Behavioral: Healthy Aging (HA) The HA group will receive a health education intervention based on topics from several sources, including the National Institute on Aging's Age Pages, University of Pittsburgh's 10 Keys to Healthy Aging; and Stanford University's Successful Aging program, among other topics . The HA intervention will receive ongoing staff contact, and will provide participants with excellent information on health-related topics. Biweekly 45-minute lectures will be given during months 1 to 6, and once per month during months 7 to 9. After each session, participants will engage in a 15-minute stretching routine. During months 10 to 12, no lectures will be given. After completion of the 12-month assessments, participants will receive a 12-month membership to the YMCA at no cost.
  Interventions: Other: Healthy Aging (HA)

INTERVENTIONS:
Behavioral: Prosocial Behavior Physical Activity (PBPA) — The PBPA condition involves a cognitive-behavioral intervention to teach participants the behavioral skills to engage in independent physical activity. Participants will engage in supervised physical activity delivered two times a week during months 1 to 3 at the William G. White, Jr. Family YMCA in Winston-Salem, NC. During months 4 to 6, supervised sessions will be held once per week, and sessions will be held once per month in months 7 to 9. Participants will engage in completely independent physical activity in months 10 to 12. PBPA participants will also be able to earn boxes of food for donation to the Second Harvest Food Bank (SHFB) of Northwest North Carolina based upon their weekly physical activity. Lowe's Foods, a regional grocery chain, will donate the food. Participants in the PBPA intervention also will receive a 12-month membership to the William G. White, Jr. Family YMCA at no cost.
  Arms: Prosocial Behavior Physical Activity
Other: Healthy Aging (HA) — The HA group will receive a health education intervention based on topics from several sources, including the National Institute on Aging's Age Pages, University of Pittsburgh's 10 Keys to Healthy Aging; and Stanford University's Successful Aging program, among other topics . The HA intervention will receive ongoing staff contact, and will provide participants with excellent information on health-related topics. Biweekly 45-minute lectures will be given during months 1 to 6, and once per month during months 7 to 9. After each session, participants will engage in a 15-minute stretching routine. During months 10 to 12, no lectures will be given. After completion of the 12-month assessments, participants will receive a 12-month membership to the YMCA at no cost.
  Arms: Healthy Aging (HA)

SUMMARY:
The purpose of this 12-month study is to compare how well two programs help older adults make physical activity a regular habit.

DETAILED DESCRIPTION:
Although only a small percentage of older adults engage in habitual physical activity, previous studies have demonstrated interventions that include cognitive-behavioral strategies can enhance long-term, independent physical activity. In addition, there are episodic charity events, such as charity walks, that attract large numbers of participants of all age ranges to engage in moderate-intensity physical activity. These actions are a form of prosocial behavior, defined as voluntary, intentional behavior that results in benefits for another. The opportunity to help others seems to be a motive in inspiring these individuals to at least engage in one session of moderate physical activity. Thus, the current research project contemplates whether prosocial behavior may be implemented as a viable behavioral incentive for long-term physical activity.

Participants in the Prosocial Behavior Physical Activity (PBPA) intervention will receive a cognitive-behavioral intervention to teach participants the behavioral skills necessary to engage in long-term (12-month) independent physical activity. Participants in the Healthy Aging (HA) intervention will receive excellent educational sessions based on a number of topics of relevance to older adults. Both programs will provide supervised stretching sessions so that participants learn how to safely and effectively improve flexibility, which helps reduce the likelihood of falls and disability. However, the PBPA intervention will also allow participants to earn food for donation to Second Harvest Food Bank based on their regular physical activity and volunteer time.

ELIGIBILITY:
Inclusion Criteria:

* age 55 years or older
* physically underactive
* no evidence of any major psychological illness
* residence within 20 miles of study site
* plans to remain in area for duration of study

Exclusion Criteria:

* currently engaging in regular physical activity
* self-reported evidence of cardiovascular disease
* self-reported evidence of diabetes
* self-reported falling within the past year
* alcohol consumption greater than 14 drinks per week
* inability to understand English
* plans to move from area
* participation in another medical intervention study
* severe hearing or sight impairments

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
physical activity | 12 months
  Self-reported physical activity will be assessed using a questionnaire at 4 time points among all participants; (1) at baseline before randomization; (2) 3 months after the interventions begin; (3) 6 months after the interventions begin; and (4) 12 months after the interventions begin

SECONDARY OUTCOMES:
physical function | 12 months
  A series of 3 physical function tests will be administered to all participants at three time points: (1) at baseline before randomization; (2) 3 months after the interventions begin; and (3) 12 months after the interventions begin. All of the tests are brief and uncomplicated to perform.

CONTACTS AND LOCATIONS:
Overall Officials: Capri G Foy, Ph.D., Principal Investigator — Wake Forest University Baptist Health
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Foy CG, Vitolins MZ, Case LD, Harris SJ, Massa-Fanale C, Hopley RJ, Gardner L, Rudiger N, Yamamoto K, Swain B, Goff DC Jr, Danhauer SC, Booth D, Gaspari J. Incorporating prosocial behavior to promote physical activity in older adults: rationale and design of the Program for Active Aging and Community Engagement (PACE). Contemp Clin Trials. 2013 Sep;36(1):284-97. doi: 10.1016/j.cct.2013.07.004. Epub 2013 Jul 19. PMID 23876672
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568